CLINICAL TRIAL: NCT06017986
Title: Metabolic and Physiological Effects of Processing on Food Reward Encoding
Brief Title: The Effect of Processing on Food Reward
Acronym: PFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Alexandra DiFeliceantonio, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-1052
Record Dates: First submitted 2023-08-01; First posted 2023-08-30 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Stimulus: UPF1 (Experimental): In a whole room metabolic chamber participants will consume a ~300 kcal meal consisting of ultra-processed foods as determined by the widely used NOVA scale. The whole room metabolic chamber will allow for collection of simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). Measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial).
  Interventions: Other: Ultra-processed food - Picture Set Meal; Other: Ultra-processed food - Additives Meal; Other: Ultra-processed food - Ingredients Meal; Other: Minimally Processed Food - Picture Set Meal; Other: Minimally Processed Food - Additives Meal; Other: Minimally Processed Food - Ingredients Meal
- Stimulus: UPF2 (Experimental): In a whole room metabolic chamber participants will consume a ~300 kcal meal consisting of ultra-processed foods as determined by the widely used NOVA scale. The whole room metabolic chamber will allow for collection of simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). Measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial).
  Interventions: Other: Ultra-processed food - Picture Set Meal; Other: Ultra-processed food - Additives Meal; Other: Ultra-processed food - Ingredients Meal; Other: Minimally Processed Food - Picture Set Meal; Other: Minimally Processed Food - Additives Meal; Other: Minimally Processed Food - Ingredients Meal
- Stimulus: UPF3 (Experimental): In a whole room metabolic chamber participants will consume a ~300 kcal meal consisting of ultra-processed foods as determined by the widely used NOVA scale. The whole room metabolic chamber will allow for collection of simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). Measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial).
  Interventions: Other: Ultra-processed food - Picture Set Meal; Other: Ultra-processed food - Additives Meal; Other: Ultra-processed food - Ingredients Meal; Other: Minimally Processed Food - Picture Set Meal; Other: Minimally Processed Food - Additives Meal; Other: Minimally Processed Food - Ingredients Meal
- Stimulus: MPF1 (Active Comparator): In a whole room metabolic chamber participants will consume a ~300 kcal meal consisting of minimally processed foods as determined by the widely used NOVA scale. The whole room metabolic chamber will allow for collection of simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). Measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial).
  Interventions: Other: Ultra-processed food - Picture Set Meal; Other: Ultra-processed food - Additives Meal; Other: Ultra-processed food - Ingredients Meal; Other: Minimally Processed Food - Picture Set Meal; Other: Minimally Processed Food - Additives Meal; Other: Minimally Processed Food - Ingredients Meal
- Stimulus: MPF2 (Active Comparator): In a whole room metabolic chamber participants will consume a ~300 kcal meal consisting of minimally processed foods as determined by the widely used NOVA scale. The whole room metabolic chamber will allow for collection of simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). Measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial).
  Interventions: Other: Ultra-processed food - Picture Set Meal; Other: Ultra-processed food - Additives Meal; Other: Ultra-processed food - Ingredients Meal; Other: Minimally Processed Food - Picture Set Meal; Other: Minimally Processed Food - Additives Meal; Other: Minimally Processed Food - Ingredients Meal
- Stimulus: MPF3 (Active Comparator): In a whole room metabolic chamber participants will consume a ~300 kcal meal consisting of minimally processed foods as determined by the widely used NOVA scale. The whole room metabolic chamber will allow for collection of simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). Measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial).
  Interventions: Other: Ultra-processed food - Picture Set Meal; Other: Ultra-processed food - Additives Meal; Other: Ultra-processed food - Ingredients Meal; Other: Minimally Processed Food - Picture Set Meal; Other: Minimally Processed Food - Additives Meal; Other: Minimally Processed Food - Ingredients Meal

INTERVENTIONS:
Other: Ultra-processed food - Picture Set Meal — A meal containing ultra-processed foods derived from the picture set used in the Becker-Degroot-Marschak auction paradigm.
Other: Ultra-processed food - Additives Meal — A meal containing ultra-processed foods that very on degree of additives.
Other: Ultra-processed food - Ingredients Meal — a meal containing ultra-processed foods that very on degree of processing but not ingredients.
Other: Minimally Processed Food - Picture Set Meal — a meal containing minimally processed foods derived from the picture set used in the Becker-Degroot-Marschak auction paradigm.
Other: Minimally Processed Food - Additives Meal — A meal containing minimally processed foods that very on degree of additives.
Other: Minimally Processed Food - Ingredients Meal — A meal containing minimally processed foods that very on degree of processing but not ingredients.

SUMMARY:
The minimally processed diets of our ancestors have been rapidly replaced by UPFs driving poor diet to become the leading risk factor for preventable death globally. Hence, it is essential to understand what properties of UPF are driving their overconsumption to reduce diet-related mortality. To address this gap in knowledge this proposal will test:

* If UPFs have a greater post meal metabolic response when compared to MPFs an essential signal for food reward
* Through the use of an auction task paradigm if UPFs overvalued and if this value is differentially encoded in the brain This study is a fully cross-over design in that each participant receives all conditions and therefore serves as their own control. All orders of foods will be counterbalanced. Although participants cannot be blinded to the conditions as they must be aware of the foods they are eating, they will not be made aware that the key manipulation is food processing. On different days participants will come to the lab and consume a meal containing either minimally or ultra-processed foods as determined by the widely used NOVA (not an acronym) scale. These conditions will be consumed in a whole room metabolic chamber allowing for simultaneous measurement of multiple metabolic responses (glucose, insulin, and metabolic rate). These measures will be collected for 45 min before consumption of the meal (baseline) and for 3 hours after consumption (post-prandial). All participants will also undergo a Becker-Degroot-Marschak auction paradigm that consists of foods that are either minimally or Ultra-processed in the MRI scanner. Food value will be measure in participants' willingness to pay for each food and Neural responses will be measured during presentation of the food cues.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-24.9 kg/m2
* Not pregnant or planning to become pregnant during study participation Residing in the Roanoke area and/or willing/able to attend sessions at the Fralin Biomedical Research Institute
* Able to speak and write in English
* Participants must be able to see a computer display clearly with or without vision correction (eyeglasses, contacts).

Exclusion Criteria:

* Claustrophobia (this would make lying in an MRI scanner or indirect calorimetry canopy very uncomfortable).

  2. History of head injury resulting in loss of consciousness for more than 10 minutes 3. Current or past diagnosis of diabetes or metabolic disorder (thyroid disease, etc.) 4. Contraindications to MRI: Individuals with pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.

  5. History of alcohol or drug dependence 6. Active neurologic disorder 8. Diagnosed eating disorder 9. Food allergies or restrictive diet

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose response to level of food processing | Immediately post intervention
  Blood glucose concentration will be assessed at baseline and at set time points for 3 hours after consumption of each condition on different days.
Blood insulin response to level of food processing | Immediately post intervention
  Blood insulin concentration will be assessed at baseline and at set time points for 3 hours after consumption of each condition on different days.
Energy expenditure in response to level of food processing | Immediately post intervention
  Whole room indirect calorimetry will be used to determine energy expenditure at baseline (for 45 minutes) and for 3 hours after consumption of each condition on different days.
Respiratory exchange ratio in response to level of food processing | Immediately post intervention
  Whole room indirect calorimetry will be used to determine respiratory exchange ratio at baseline (for 45 minutes) and for 3 hours after consumption of each condition on different days.
Substrate oxidation in response to level of food processing | Immediately post intervention
  Whole room indirect calorimetry will be used to determine substrate oxidation at baseline (for 45 minutes) and for 3 hours after consumption of each condition on different days.
Effect of food processing on food value and encoding | through study completion, an average of 3 weeks
  A food picture set of 28 that are matched on 23 visual, perceptual, and nutritional properties but vary on degree of NOVA food processing level will be used in a Becker-Degroot-Marschak auction paradigm to assess participants' brain reward response for each food.

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No